CLINICAL TRIAL: NCT04518137
Title: An Open-Label, Single-Arm Basket Study of ATG-008 for the Treatment of Patients With Advanced Solid Tumors Harboring NFE2L2, STK11, RICTOR or Other Specific Genetic Alterations
Brief Title: A Study of Evaluating the Safety and Efficacy of ATG-008 for Advanced Solid Tumors (BUNCH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the low popularity of NGS testing in China and the small number of target subjects, our company decided to adjust the research and development strategy, terminate this study and not apply for new drug registration after careful consideration.
Sponsor: Shanghai Antengene Corporation Limited (Industry)
Responsible Party: Sponsor
Organization: Antengene Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-008-AST-001
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATG-008 (Experimental): Enrolled patients will be treated with ATG-008 at an oral fixed milligram (mg) dose of 30 mg QD
  Interventions: Drug: ATG-008 30 mg, orally, QD, each 4 week (28-day) a cycle

INTERVENTIONS:
Drug: ATG-008 30 mg, orally, QD, each 4 week (28-day) a cycle — 48 patients enrolled will be treated with 30mg QD of ATG-008, orally, each 4 week (28-day) a cycle
  Other Names: ATG-008

SUMMARY:
This is a single-arm and open-label study of ATG-008 for the Treatment of Patients With advanced Solid Tumors harboring NFE 2L2, STK11, RICTOR or other specific genetic alterationts

DETAILED DESCRIPTION:
This is a single-arm and open-label study. Approximately 10-12 patients will be enrolled per each genetic alterration group in the study. ATG-008 is the monotherapy for advanced solid tumors with 30mg QD. The clinical efficacy, safety and tolerability of ATG-008 will be evaluated. Addtionalal dose levels may apply after the efficacy/safety and tolerabitly of 30mg QD has been accessed by Sponosor and study steering committee.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and provide informed consent.
2. Males or females of 18 years of age or older
3. Have histologically-proven measurable, or evaluable advanced (systemically or locally progressive), or metastatic solid tumors or the locally advanced disease is not amenable to local therapy, who have failed, or are intolerant to standard therapy or for whom no standard therapy is available. (For subjects with hepatocellular carcinoma, the diagnosis needs to be supported by dynamic computed tomography [CT]/magnetic resonance imaging, if pathological confirmation is not attainable) and agree to provide tumor tissues (within 24 months) for genomic analysis (For subjects who can provide the first NGS reports[The report was based on tumor tissues within 12 months prior to the subject's test] within 12 months prior to screening and has target gene variation(s), it is recommended to provide their tumor tissue samples to the central laboratory for testing, but the test results will not affect the inclusion/exclusion evaluation of the subjects).
4. Harboring with below specific genetic alterations:

   1. NFE2L2 mutations
   2. STK11 mututions
   3. RICTOR amplifications
   4. Other genetic alterations maybe enrolled after discussion with Sponsor medical monitor
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. A life expectancy longer than 3 months in the opinion of the Investigator.
7. Adequate hematologic functions, as defined by: absolute neutrophil counts ≥ 1500/mm3; a hemoglobin level ≥ 9 g/dL; a platelet count ≥ 100,000/mm3.
8. Adequate hepatic function defined by: a total bilirubin level ≤ 1.5 × of upper limit of normal (ULN); aspartate transaminase and alanine transaminase levels ≤ 2.5 × ULN(AST and ALT ≤5 × ULN for subjects with liver metastasis).
9. Adequate renal function, as defined by the creatinine clearance ≥ 50 mL/minute (as calculated by the Cockcroft-Gault formula).
10. Females of child-bearing potential must have a negative pregnancy test upon entry into this study and must be willing to use highly effective birth control upon enrollment, during the Treatment Phase and for 180 days following the last dose of study drug. A female is considered of child-bearing potential following menarche and until becoming postmenopausal (no menstrual period for a minimum of 12 months) unless permanently sterile (undergone a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).
11. If male, must be surgically sterile or willing to use highly effective birth control upon enrollment, during the Treatment Phase, and for 180 days following the last dose of study drug.
12. Child-pugh score of A or B7 (for subjects with hepatocellular carcinoma only).

Exclusion Criteria:

1. Except for hearing loss and hair loss, all toxicity from previous antitumor therapy was not recovered to≤Grade 1 (according to National Cancer Institute-Common Terminology Criteria Adverse Events [NCI-CTCAE], version 5.0).
2. Concurrent unstable or uncontrolled medical conditions, including:

   1. Active systemic infections;
   2. Poorly controlled hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg), or poor compliance with antihypertensive agents;
   3. Clinically significant arrhythmia, unstable angina pectoris, congestive heart failure (Class II or IV of New York Heart Association) or acute myocardial infarction;
   4. Uncontrolled diabetes or poor compliance with hypoglycemic agents (as defined: HbA1c >7%);
   5. The presence of chronically unhealed wound or ulcers;
   6. Other chronic diseases, which, in the opinion of the Investigator, could compromise safety of the patient or the integrity of the study.
3. Poorly controlled pleural effusion or pericardial effusion (with clinical symptoms, fluctuating or repeated drainage of effusion, oral diuretics, etc) existed in the screening period. During the screening period, there are ascites that can be detected on physical examination, or clinical symptoms caused by ascites, or special treatment is required, such as repeated drainage, intraperitoneal drug perfusion, etc (the presence of a small amount of ascites that can only be detected by imaging examination may be considered for enrollment).
4. CNS metastases or involvement (except for the subjects with stable symptoms and no recurrence within 2 years and be likely to obtain benefit from the study determined by the investigator).
5. History of hepatic encephalopathy (only applicable to hepatocellular carcinoma subjects).
6. Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix. (Subjects with a previous malignancy but without evidence of disease for ≥ 5 years can participate).
7. Females who are pregnant, lactating, or intend to become pregnant during their participation in this study.
8. Current or prior use of immunosuppressive medication within 14 days before the first dose. The following are exceptions to this criterion:

   1. Intranasal, inhaled, topical steroids or local steroid injections (eg, intra-articular injection), OR
   2. systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent, OR
   3. steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
9. Unable to swallow ATG-008 tables.
10. Major surgery was performed within 28 days prior to screening.
11. Had anti-tumor therapy (including radiotherapy and interventional therapy, etc), systemic chemotherapy, hormone regulation therapy (such as tamoxifen), traditional Chinese medicine therapy with anti-tumor indications, or clinical trial drugs, and medical devices within 28 days prior to screening.
12. History of primary immunodeficiency or allogeneic transplantation.
13. History of human immunodeficiency virus (HIV) infection and/or acquired immunodeficiency syndrome.
14. Active hepatitis B (HBsAg active), active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV RNA test at Screening.
15. History of interstitial lung disease.
16. Receipt of live attenuated vaccines within 30 days prior to screening. Subjects, if enrolled, should not receive live or live attenuated vaccines during the study.
17. Use/eating of drugs or food known to have potent CYP3A4 inhibitory effects within 2 weeks prior to screening, including but not limited to, atazanavir, clarithromycin, Indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, vinegar oleandomycin, voriconazole, grapefruit and grapefruit juice.
18. Use of drugs known to have strong CYP3A4 induction within 2 weeks prior to screening, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampicin, and St. John's wort.
19. Use of drugs as CYP3A4 substrates (with stenosis treatment index) within 2 weeks prior to screening, including but not limited to dihydroergodemine, ergodemine, pimozide, astimidazole, cisapride, and terfenadine.
20. Treatment with mTOR（TORC1and/orTORC2）inhibitor, included but not limited to sirolimus, temsirolimus, everolimus, and other experimental or approved mTOR/PI3K/AKT inhibitors.
21. The subject is the investigator, sub-investigator, or anyone directly involved in the conduct of the study.
22. The investigator considers that complications or other conditions of the subject may affect the compliance with the protocol or make the subject unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
ORR | 19 months
  Percentage of subjects with PR, or CR

SECONDARY OUTCOMES:
DOR | 19 months
  Duration of time from first occurrence of CR or PR until the first date that disease progression is objectively documented
DCR | 19 months
  Proportion of patients who achieve CR, PR, or SD for a minimum of 4 weeks, following the first dose of study drug (i.e., CR+PR+SD)
OS | 19 months
  Duration of time from the first dose of study drug until death due to any cause
PFS | 19 months
  Duration of time from the first dose of study drug until progression or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD; PhD, Principal Investigator — Chinese Academay of Medical Science and Peking Union Medical College
Locations (4):
- China (4):
  - National Cancer Center/Cancer Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality
  - Chongqing university cancer hospital, Chongqing, Chongqing Municipality
  - The first affiliated hospital of xiamen university, Xiamen, Fujian
  - West China Hospital of Sichuan University, Chengdu, Sichuan